CLINICAL TRIAL: NCT06152900
Title: Clinical Evaluation of the Safety and Efficacy of Electronic Stimulation for Non-Invasive Circumferential Reduction and Muscle Toning
Brief Title: Safety and Efficacy of Electronic Stimulation for Circumferential Reduction and Muscle Toning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CynosureLutronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFL19006
Record Dates: First submitted 2023-11-22; First posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Fat Necrosis; Muscle Stimulation
MeSH Terms: conditions — Fat Necrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment Arm (Experimental): All subjects enrolled in the study will be placed into the treatment arm of the study, to be treated by the Accufit device.
  Interventions: Device: Accufit

INTERVENTIONS:
Device: Accufit — Magnet-based and Direct muscle stimulation devices are commonly used to generate current flow through the muscles in order to activate the muscle. The Accufit Electrical Muscle Stimulation device is an FDA cleared device having a two-channel stimulator that provides up to 8 electrodes with waveforms of interferential and biphasic for muscle stimulation. The Accufit system is indicated for relaxation of muscles, muscle re-education, reduction of pain and increased local blood circulation.
  Muscle stimulation technology has been around for many decades and has been shown to be safe and effective for a variety of clinical applications. The foundational basis for the technology revolves around electrical current flowing through the muscle can be used to activate the muscle.
  Other Names: ME Sys*STIM 240

SUMMARY:
Open-label, baseline-controlled, multi-center study evaluating an electrical muscle stimulation system for circumferential reduction and muscle toning. The study will enroll up to 100 subjects desiring circumferential reduction and muscle toning. Each subject will receive up to 12 bi-weekly treatments over a 6-week period. Follow Up Visits planned for 2, 30- and 90-days post treatment. Measurement outcomes will be compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand and voluntarily provide written informed consent.
2. Healthy male or female, ≥ 18 years to 65 years of age seeking treatment for improved muscle strength and muscle toning in their core and extremities.
3. Subject is determined to be physically fit and agrees to not making any major changes in their diet or lifestyle during the study.
4. Able and willing to comply with the treatment/follow-up schedule and requirements.
5. Women of child-bearing age are required to be using a reliable method of birth control at least 3 months prior to study enrollment and for the duration of the study as well as have a negative Urine Pregnancy test at baseline.

Exclusion Criteria:

1. Pregnant in the last 3 months, intending to become pregnant, postpartum or nursing in the last 6 months.
2. Any previous liposuction/lipo-sculpture or any type of surgical procedure in the treatment area in the past 12 months.
3. History of immunosuppression/immune deficiency disorders (including AIDS and HIV infection) or use of immunosuppressive medications, 6 months prior to and during the study.
4. History of hyperlipidemia, diabetes mellitus, hepatitis, blood coagulopathy or excessive bleeding.
5. Having a history of skin cancer or any other cancer in the areas to be treated, including presence of malignant or premalignant pigmented lesions.
6. Having a permanent implant in the treatment area such as metal plates or an injected chemical substance such as silicone in the treatment area.
7. Suffering from significant skin conditions in the treatment area or inflammatory skin conditions including but not limited to open lacerations, abrasions, herpes sores, cold sores, active infections.
8. Poor skin quality (severe laxity).
9. Abdominal wall, muscular abnormality or hernia on physical examination.
10. As per the investigator's discretion, any physical or mental condition which may make it unsafe for the subject to participate.
11. Subjects unwilling or unable to adhere to all study requirements for treatment and follow-up.
12. Investigator may exclude any subject at any time at his/her discretion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Photographic Evaluation | Baseline, 48-hours post treatment, 30-day FU, 90-day FU
  Photographic evaluation by an independent, blinded reviewer with correct identification of pre-treatment baseline images when compared to post-treatment images taken at follow up visits (48 hours, 30 days, 90 days).Results will be reported as a % of the correctly identified post treatment photographs chosen per Blinded Reviewer. An average of the % of the correctly identified post treatment photographs chosen by Blinded Reviewer will be calculated and used to determine efficacy.

SECONDARY OUTCOMES:
Circumferential Reduction | Baseline, 30-day FU, 90-day FU
  Reduction in circumference as measured by Seca Circumferential System at follow up visits compared to baseline measurement. Measurements were taken of the right and left arm in both a relaxed and engaged position.
Subject Satisfaction | 30-day FU, 90-day FU
  Assess subject satisfaction using Satisfaction survey at each follow up visit. Scores available in the scale include the following:
  1. - Very Satisfied
  2. - Satisfied
  3. - Neutral
  4. - Dissatisfied
Global Aesthetic Improvement Scale | 30-day FU, 90-day FU
  A scale to assess the overall improvement in a subject's condition in an unblinded fashion. Choices on the scale include the following:
  1. - Very Much Improved
  2. - very Improved
  3. - Improved
  4. - No Change
  5. - Worsened
Muscle Strength | Baseline, 30-day FU, 90-day FU
  Improvement in muscle strength of the treated extremity as measured by a dynamometer at follow up visits compared to baseline measurements. Subjects are asked to hold onto a handheld device which will then be used to measure the strength of the bicep and tricep muscles.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Lutronic US Headquarters, Billerica, Massachusetts
  - Union Square Dermatology, New York, New York

IPD SHARING:
Plan to Share IPD: No
No IPD Sharing planned at this time.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-08): https://cdn.clinicaltrials.gov/large-docs/00/NCT06152900/Prot_SAP_000.pdf